CLINICAL TRIAL: NCT03668535
Title: Filling of the Urinary Bladder During Difficult Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammad Abdel-Rahman Mohammad Ahmed, Doctor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OBGYN 004
Record Dates: First submitted 2018-09-09; First posted 2018-09-12 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Urinary Tract Injury; Cesarean Section Complications
Keywords: Urinary; Bladder; Injury; Cesarean
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Two groups of women with difficult Cesarean Section at risk of urinary bladder injury. Group A will receive the intervention. Group B will not receive the intervention.
Who Masked: Participant, Investigator
Masking Description: closed envelop will be used for randomization. The patient and the investigator will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bladder Filling arm (Active Comparator): Group A have triple-way urethral catheter insertion before establishment of anaesthesia. Evaluation of the drained urine is done (including: amount, character, and simple for culture and sensitivity). Instillation of 200 ml sterile saline is done by 50 ml syringe through the irrigation way. The irrigation way is closed temporarily by artery forceps. After laparotomy the bladder may be deflated by 50 ml or further inflated by 50 ml if needed to allow comfortable dissection.
  Interventions: Procedure: Bladder Filling
- Bladder deflation arm (Active Comparator): Group B have Foley's catheter is inserted as usual. The catheter is connected freely to urinary bag.
  Interventions: Procedure: Bladder deflation

INTERVENTIONS:
Procedure: Bladder Filling — Group A have a triple-way urethral catheter insertion before establishment of anaesthesia. Evaluation of the drained urine is done (including: amount, character, and simple for culture and sensitivity). Instillation of 200 ml sterile saline is done by 50 ml syringe through the irrigation way. The irrigation way is closed temporarily by artery forceps. After laparotomy the bladder may be deflated by 50 ml or further inflated by 50 ml if needed to allow comfortable dissection.
  Arms: Bladder Filling arm
Procedure: Bladder deflation — Group B have Foley's catheter is inserted as usual. The catheter is connected freely to urinary bag.
  Arms: Bladder deflation arm

SUMMARY:
Risk factors for bladder injury during Cesarean Section are well known. Most of cases of bladder injury occur in presence of previous Cesarean Sections, morbidly adherent placenta, or previous bladder injury. limited evidence suggest that bladder filling may decrease the incidence of bladder injury. n our study, we compared the outcome of urinary bladder filling during Cesarean Section in cases at high risk of bladder injury.

DETAILED DESCRIPTION:
In women at risk of bladder injury, such as in presence of previous Cesarean Section(s), there may tough adhesions between the bladder and the lower uterine segment. Trial of separation of the bladder in such circumstances may result in bladder injury. Filling of the bladder will delineate the contour of the bladder and clarify the proper plane of dissection. In a recent randomized clinical trial lower bladder filling resulted in non-significant decrease in the rate of bladder injury in women with placenta percreta. In our study, we compared the outcome of urinary bladder filling during Cesarean Section in cases at high risk of bladder injury.

Patients and Methods Inclusion criteria: Pregnant women at gestation from 20- 41 weeks who have any of the following risk factors

1. Previous Cesarean Section 3 times or more
2. Previous history of bladder injury during Cesarean Section
3. Operative report of extensive adhesions in the last Cesarean Section
4. Cesarean Section for placenta accreta spectrum Methods This is a randomized controlled trial done at the department of Obstetrics & Gynaecology unit, South Valley University from August 1st, 2017until the 30th of August 2018. The research is approved by the Committee of Ethics for Biomedical Researches, South Valley University at June 2017. All cases have informed consent before inclusion in the research. Closed envelop is used to randomized patients to either group. Group A: are cases of Cesarean section who have the intervention. Group: are cases of Cesarean section who do not have the intervention.

The intervention:

Triple-way urethral catheter insertion before establishment of anaesthesia. Evaluation of the drained urine is done (including: amount, character, and simple for culture and sensitivity). Instillation of 200 ml sterile saline is done by 50 ml syringe through the irrigation way. The irrigation way is closed temporarily by artery forceps. After laparotomy the bladder may be deflated by 50 ml or further inflated by 50 ml if needed to allow comfortable dissection. All Cesarean sections in both groups are done by the same surgeon supported by the same team in the same hospital. The Cesarean sections are done under spinal or general anaesthesia through pfannenstiel's incision. The catheter is removed 12 hours after Cesarean section. Postoperative follow up is maintained until 3 months from the time of the Cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Previous Cesarean Section 3 times or more
* Previous history of bladder injury during Cesarean Section
* Operative report of extensive adhesions in the last Cesarean Section
* Cesarean Section for placenta accreta spectrum

Exclusion Criteria:

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women undergoing Cesarean Section
Enrollment: 266 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
bladder injury | 3 months
  the intra-operative rate of urinary bladder injury

SECONDARY OUTCOMES:
Operative time | 3 months
  Operative time in minutes
post-operative voiding dysfunction | 3 months
  post-operative voiding dysfunction in the form of dysuria or retention
operative blood loss | 3 months
  estimated blood loss in mL
Urinary bladder fistulae | 3 months
  development of bladder fistulae

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad AM Ahmed, MD, Principal Investigator — South Valley University, Qena Faculty of Medicine, Obstetrics and Gynecology Department, Qena, Qena, Egypt
Locations (1):
- South Valley University, Qena Faculty of Medicine, Obstetrics and Gynecology Department, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared in unanonomous manner with the predetermined group of researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: throughout the period of research until end of the study
Access Criteria: IPD will be shared with the predetermined group of researchers as accepted by the local ethical and research committee.

REFERENCES:
- [Background] Salman L, Aharony S, Shmueli A, Wiznitzer A, Chen R, Gabbay-Benziv R. Urinary bladder injury during cesarean delivery: Maternal outcome from a contemporary large case series. Eur J Obstet Gynecol Reprod Biol. 2017 Jun;213:26-30. doi: 10.1016/j.ejogrb.2017.04.007. Epub 2017 Apr 5. PMID 28411456
- [Background] Alanwar A, Al-Sayed HM, Ibrahim AM, Elkotb AM, Abdelshafy A, Abdelhadi R, Abbas AM, Abdelmenam HS, Fares T, Nossair W, Abdallah AA, Sabaa H, Nawara M. Urinary tract injuries during cesarean section in patients with morbid placental adherence: retrospective cohort study. J Matern Fetal Neonatal Med. 2019 May;32(9):1461-1467. doi: 10.1080/14767058.2017.1408069. Epub 2017 Dec 3. PMID 29157027
- [Background] Pandey D, Mehta S, Grover A, Goel N. Indwelling Catheterization in Caesarean Section: Time To Retire It! J Clin Diagn Res. 2015 Sep;9(9):QC01-4. doi: 10.7860/JCDR/2015/13495.6415. Epub 2015 Sep 1. PMID 26500959
- [Background] Senanayake H. Elective cesarean section without urethral catheterization. J Obstet Gynaecol Res. 2005 Feb;31(1):32-7. doi: 10.1111/j.1447-0756.2005.00237.x. PMID 15669989
- [Background] Acharya S, Uprety DK, Pokharel HP, Amatya R, Rai R. Cesarean section without urethral catheterization: a randomized control trial. Kathmandu Univ Med J (KUMJ). 2012 Apr-Jun;10(38):18-22. doi: 10.3126/kumj.v10i2.7337. PMID 23132469
- [Background] Abdel-Aleem H, Aboelnasr MF, Jayousi TM, Habib FA. Indwelling bladder catheterisation as part of intraoperative and postoperative care for caesarean section. Cochrane Database Syst Rev. 2014 Apr 11;2014(4):CD010322. doi: 10.1002/14651858.CD010322.pub2. PMID 24729285
- [Background] Ozcan HC, Balat O, Ugur MG, Sucu S, Tepe NB, Kazaz TG. Use of Bladder Filling to Prevent Urinary System Complications in the Management of Placenta Percreta: a Randomized Prospective Study. Geburtshilfe Frauenheilkd. 2018 Feb;78(2):173-178. doi: 10.1055/s-0044-100039. Epub 2018 Feb 19. PMID 29479114
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246